CLINICAL TRIAL: NCT04504305
Title: A Double-blind, Randomized, Placebo-controlled Study to Assess the Efficacy of Investigational Product Nerve Support Formula on the Neuropathic Pain in Individuals Suffering From Type II Diabetes Mellitus.
Brief Title: To Assess the Efficacy of Investigational Product on the Neuropathic Pain in Individuals Suffering From Type II Diabetes Mellitus.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VC/190403/NUEROPAWAY/PN
Record Dates: First submitted 2020-08-04; First posted 2020-08-07 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2020-08

CONDITIONS: Diabetic Neuropathies; Insomnia Due to Medical Condition
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuropaway (Active Comparator)
  Interventions: Other: NeuropAWAY
- Microcystalline cellulose (Placebo Comparator)
  Interventions: Other: Microcystalline cellulose

INTERVENTIONS:
Other: NeuropAWAY — 2 capsules thrice daily to be taken half an hour prior to meal.
  Arms: Neuropaway
Other: Microcystalline cellulose — 2 capsules thrice daily to be taken half an hour prior to meal.
  Arms: Microcystalline cellulose

SUMMARY:
this study is to be carried out to examine the effect of Investigation product on diabetic individuals suffering from diabetic neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Male and Females aged ≥ 40 and ≤ 65 years of age.
* Participants with primary complaints of lower limb pain.
* History of Diabetes mellitus for more than one year.
* Participants with HbA1c ≥ 7.1 and ≤ 9.5%

Exclusion Criteria:

* Diagnosed with severe cardiac disease
* Uncontrolled hypertension defined as systolic blood pressure ≥ 139 and diastolic blood pressure ≥ 85.
* Type II DM with history of foot ulcers in the last six months prior to the study
* History of nerve damage not due to Painful Diabetic Neuropathy.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
effect of investigational product on diabetic individual suffering from diabetic neuropathy assessed by 11 point numeric rating scale. | 42 days
  pain intensity will be assessed by 11 point numeric rating scale where 0 indicates no pain and 10 indicates worst possible pain

SECONDARY OUTCOMES:
effect of investigational product on diabetic individual suffering from diabetic neuropathy assessed by Brief pain inventory. | 42 days
effect of investigational product on diabetic individual suffering from diabetic neuropathy assessed by insomnia Severity index. | 42 Days
effect of investigational product on diabetic individual suffering from diabetic neuropathy assessed by Neuropathy total symptom score - 6 . | 42 Days

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Stress Test Clinic, Mumbai, Maharashtra
  - Shantaee, Mumbai, Maharashtra